CLINICAL TRIAL: NCT06662591
Title: A Multi-Center Multi-Omics Approach for Investigating Genetic and Epigenetic Mechanisms in Autism Spectrum Disorder
Brief Title: Investigation of the Genetic and Environmental Causes of Autism: a Multi-Center Study
Acronym: ASD-Omics-TR
Status: Not yet recruiting | Type: Observational
Sponsor: Research and Treatment Society of Genetic Disorders (Other)
Collaborators: İnvitrotek A.Ş. (Unknown); Selcuk University (Other); Istanbul Cerrahpasa Faculty of Medicine, Department of Child and Adolescent Psychiatry (Unknown); Istanbul Medeniyet University Faculty of Medicine, Department of Child and Adolescent Psychiatry (Unknown); Ankara SBÜ Gülhane Faculty of Medicine, Department of Child and Adolescent Psychiatry (Unknown); Ankara Gazi Faculty of Medicine, Department of Child and Adolescent Psychiatry (Unknown); Izmir Katip Çelebi Faculty of Medicine, Department of Child and Adolescent Psychiatry (Unknown); Şanlıurfa Harran University Faculty of Medicine, Department of Child and Adolescent Psychiatry (Unknown); Erzurum Atatürk University Faculty of Medicine, Department of Child and Adolescent Psychiatry (Unknown); Trabzon Karadeniz Technical University Faculty of Medicine, Department of Child and Adolescent Psychiatry (Unknown); Denizli Pamukkale University Faculty of Medicine, Department of Child and Adolescent Psychiatry (Unknown); Gaziantep University, Department of Child and Adolescent Psychiatry (Unknown); Afyonkarahisar University of Health Sciences, Faculty of Medicine, Department of Child and Adolescent Psychiatry (Unknown); Uludag University (Other); Giresun University, Department of Child and Adolescent Psychiatry (Unknown); Baskent University (Other); Istanbul Medeniyet University, Department of Psychiatry (Unknown); Necmettin Erbakan University (Other); Istanbul Çam and Sakura City Hospital, Department of Child and Adolescent Psychiatry (Unknown)
Responsible Party: Sponsor
Other Study IDs: ERC2025SYG-TR-ASD-MultiOmics; HRU.24/16/37 (Other: Turkish Medicines and Medical Devices Agency Ethics Committee-HARRAN ÜNİVERSİTESİ KLİNİK ARAŞTIRMALAR ETİK KURULU); ERC2025SYG-TR-ASD-MultiOmics (Other: Horizon European Research Council Synergy Grants(HORIZON-ERC-SYG))
Record Dates: First submitted 2024-10-24; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Autism Spectrum Disorder (ASD)
Keywords: Autism Spectrum Disorder; Genetic Variants; Epigenetics; Transcriptomics; DNA Methylation; Gene Expression Regulation; Polygenic Risk Score; Biomarkers; Whole Genome Sequencing; Epitranscriptomics; Expression Quantitative Trait Loci; Methylation Quantitative Trait Loci; Differentially Methylated Regions; Epigenome-Wide Association Study; Genome-Wide Association Study; RNA Sequencing; Allele-Specific Methylation; Single Nucleotide Polymorphisms; Copy Number Variations; Insertions and Deletions
MeSH Terms: conditions — Autism Spectrum Disorder; Genetic Risk Score

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Biospecimen Retention: Samples With DNA — 1. Venous Blood Samples:
     Analysis: These will be used for Whole Genome Sequencing (WGS), Whole Genome Bisulfite Sequencing (WGBS) for DNA methylation analysis, and RNA-Whole Transcriptome analysis to assess gene expression.
  2. Nasal Swab Samples:
     Analysis: These will be utilized for Whole Genome Bisulfite Sequencing (WGBS) for methylation analysis and RNA-Whole Transcriptome analysis to explore tissue-specific gene expression profiles.
  3. Serum or Plasma Samples (from venous blood, Not from all case-controls):
  Analysis: These samples will be used for ELISA to quantify protein levels, such as cytokines, growth factors, or other biomarkers of interest in ASD.
  Purpose: ELISA will provide insights into the biological effects of genetic and epigenetic changes by assessing the corresponding protein expression levels in the blood.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- ASD Case Group: Represents individuals diagnosed with Autism Spectrum Disorder (ASD), who will undergo genetic, epigenetic, and transcriptomic analysis.
- Control Group: Represents unaffected individuals, serving as the comparison group for genetic and molecular analyses.
- HOT Cluster Biomarker Group: Represents participants selected after secondary outcome results based on HOT cluster analysis, who will undergo ELISA to study potential biomarkers derived from RNA transcriptome pathway analysis.

SUMMARY:
The goal of this observational study is to investigate the genetic and epigenetic mechanisms that may contribute to the development of Autism Spectrum Disorder (ASD) in individuals of different age groups. The study aims to explore how genetic variants and environmental factors interact to influence the risk of ASD.

The main questions it aims to answer are:

* Which genetic variants are most strongly associated with the development of ASD?
* How do environmental factors, such as prenatal exposure, influence these genetic risks?
* Can the combination of genetic and epigenetic data improve early detection or intervention strategies for ASD?

Participants will:

* Provide biological samples for genetic and epigenetic analysis.
* Complete detailed questionnaires regarding environmental exposures and family history.
* Participate in clinical assessments to evaluate the severity of ASD symptoms.

Researchers will compare genetic and environmental data between individuals with ASD and those without the disorder to understand how these factors may contribute to the risk of ASD. This multi-center study will take place across several universities and hospitals in Türkiye, focusing on the potential interplay between inherited genetic factors and environmental influences.

DETAILED DESCRIPTION:
Introduction to the Project The project represents an innovative, multi-center study aimed at investigating the genetic, epigenetic, and environmental underpinnings of Autism Spectrum Disorder (ASD). ASD is a complex neurodevelopmental condition that typically presents in early childhood and affects individuals in diverse ways, particularly in social communication and behavior. The disorder is marked by significant variability in symptom severity and presentation across individuals. Despite years of research, the molecular mechanisms driving the onset and progression of ASD remain elusive, making diagnosis and treatment challenging.

This research aims to fill this gap by using a multi-omics approach to better understand the biological, genetic, and environmental factors contributing to ASD. Through the integration of genomic, epigenomic, and transcriptomic data, the project seeks to uncover molecular signatures and interactions that could explain the variability in ASD presentation and severity. Additionally, the study aims to identify potential biomarkers that could lead to earlier diagnosis, better prognosis, and more personalized treatment options.

The study will be conducted across multiple research centers, with a structured and well-coordinated approach to data collection, sample processing, and analysis. This multi-disciplinary project brings together a range of expertise, including genetics, bioinformatics, clinical psychiatry, and data science, ensuring that all aspects of the research are approached with scientific rigor and precision. By analyzing samples from individuals with ASD, the project will provide new insights into the genetic and epigenetic factors involved in ASD, while also investigating the potential influence of environmental factors.

Multi-Departmental Structure and Project Integrity The project is organized into multiple specialized departments, each with a specific role in maintaining the integrity of the study and ensuring that all research activities are conducted to the highest standards. This structure allows for seamless collaboration between departments and ensures that all data is collected, processed, and analyzed with the utmost accuracy.

Overall Coordination and Oversight At the highest level, the project is managed by an overall coordinator who oversees all aspects of the research. This coordinator ensures that each department adheres to the project's goals and timeline, fostering communication between teams and facilitating the integration of clinical, genetic, and epigenetic data. Coordination ensures that any challenges arising in the course of the study are promptly addressed and that the project remains on track to meet its objectives.

The role of the overall coordinator is critical for ensuring the integration of the multi-omics data from the various research centers. The coordinator also plays a key part in the interpretation of data, working closely with the data analysis teams to ensure that the findings are cohesive and meaningful. Regular updates are shared across departments to maintain alignment with the project's overarching research goals.

Clinical Operations: Adult and Pediatric Units The clinical operations of the project are divided into two main sectors: adult and pediatric. Each sector is managed by a dedicated team that oversees clinical centers responsible for data collection. These clinical centers are located across various regions, enabling the project to gather a broad and diverse range of clinical data from individuals diagnosed with ASD.

Each clinical center follows standardized protocols for data collection, ensuring that all patient data is collected in a uniform and consistent manner. The data collection process involves the use of internationally recognized diagnostic tools, including the Autism Diagnostic Observation Schedule (ADOS) and the Social Communication Questionnaire (SCQ). These tools are essential for diagnosing ASD and for evaluating the severity of symptoms.

The clinical operations also involve the collection of sociodemographic data, developmental histories, and information on comorbid conditions. This data is gathered through questionnaires and clinical interviews conducted by trained healthcare professionals. The collection of this comprehensive dataset is critical for understanding the clinical heterogeneity of ASD and for correlating clinical symptoms with genetic and environmental data.

Genetic and Omics Divisions The genetic and omics divisions form the core of the project, providing the molecular data that will be used to uncover the genetic and epigenetic mechanisms driving ASD. The division oversees the collection, processing, and analysis of biological samples, which include venous blood and nasal swabs obtained from study participants.

Sample Collection and Processing The biological samples collected from participants undergo a rigorous and standardized process of nucleic acid extraction. This process, managed by the nucleic acid extraction and purification teams, involves isolating high-quality DNA and RNA from the blood and nasal swab samples. These samples are essential for downstream sequencing and analyses. The quality of the extracted DNA and RNA is critical, as any impurities or degradation could affect the accuracy of the genetic and epigenetic analyses.

Once extracted, the DNA and RNA samples are subjected to multiple quality control checks. These checks are overseen by the quality control and storage teams, who ensure that the nucleic acids meet the required standards for sequencing. Samples that pass the quality control checks are stored under optimal conditions, preserving their integrity until they are ready to be sequenced.

Genomic Analysis The genomic analysis of DNA samples begins with whole genome sequencing (WGS), a comprehensive technique that allows researchers to examine the entire genetic code of each participant. WGS enables the identification of a wide range of genetic variants, including single nucleotide polymorphisms (SNPs), copy number variations (CNVs), insertions and deletions (InDels), and structural variants. These variants are evaluated to determine their potential contribution to ASD.

One of the primary analyses conducted within the genomic division is the genome-wide association study (GWAS). GWAS is used to identify genetic variants that are significantly associated with ASD by comparing the frequency of variants between individuals with ASD and those without the disorder. This analysis is particularly useful for identifying common genetic variants that may contribute to ASD risk.

In addition to GWAS, the project also conducts quantitative trait locus (QTL) analysis. QTL analysis examines how genetic variants influence quantitative traits related to ASD, such as symptom severity, cognitive functioning, or developmental milestones. This type of analysis helps to elucidate the genetic basis for phenotypic variability in ASD and identifies specific variants that may contribute to differences in symptom presentation.

Epigenetic Analysis The epigenetic component of the project focuses on how environmental factors influence gene expression and contribute to the risk of ASD. DNA methylation is one of the key epigenetic mechanisms studied in this project. Using whole genome bisulfite sequencing (WGBS), researchers analyze DNA methylation patterns across the entire genome. WGBS is considered the gold standard for high-resolution DNA methylation analysis, allowing the identification of methylation changes that are associated with ASD.

Differentially methylated regions (DMRs) are genomic regions where the methylation levels differ between individuals with ASD and unaffected controls. By identifying these DMRs, researchers can pinpoint specific genomic regions where environmental factors may be influencing gene expression in individuals with ASD.

Additionally, allele-specific methylation (ASM) is explored in this study. ASM analysis investigates how methylation patterns differ between the two copies of a gene inherited from each parent. This analysis helps researchers understand how genetic and epigenetic factors interact to influence gene expression and contribute to ASD risk.

As part of the epigenetic analysis, m-QTL (methylation quantitative trait loci) analysis will be conducted to investigate the relationship between genetic variants and DNA methylation patterns across the genome. m-QTLs are genomic loci where variations in DNA sequence are associated with differences in DNA methylation levels. By identifying these loci, the project aims to uncover how genetic variation influences epigenetic regulation and, subsequently, how these interactions may contribute to the risk of developing ASD. This analysis will provide valuable insights into the interplay between genetic and epigenetic factors, helping to elucidate the molecular mechanisms that underpin ASD. Additionally, m-QTLs may serve as potential biomarkers for understanding the environmental modulation of genetic susceptibility in individuals with ASD.

The epigenetic data is also integrated with genetic data to conduct epigenome-wide association studies (EWAS). EWAS examines how DNA methylation patterns correlate with ASD, with the goal of identifying methylation marks that could serve as biomarkers for the disorder. These analyses are essential for understanding how environmental exposures, such as prenatal stress, toxins, or maternal health, may affect ASD risk through epigenetic mechanisms.

Transcriptomic Analysis The transcriptomic analysis focuses on understanding how gene expression differs between individuals with ASD and those without the disorder. RNA sequencing (RNA-seq) is used to measure the levels of gene expression in both blood and nasal swab samples. RNA-seq provides a comprehensive view of the transcriptome, which represents the complete set of RNA transcripts present in a cell or tissue at a given time.

The RNA-seq data is used to perform differential gene expression (DGE) analysis, which identifies genes that are either upregulated or downregulated in individuals with ASD. This analysis helps to uncover the molecular pathways that are disrupted in ASD and highlights potential biomarkers that could be used for early diagnosis or treatment.

In addition to identifying differentially expressed genes, the transcriptomic data is used to perform pathway analysis. Pathway analysis examines how changes in gene expression affect biological processes and cellular functions. This analysis can identify key pathways that may be disrupted in ASD, providing insights into the biological mechanisms underlying the disorder.

By comparing the gene expression profiles from both blood and nasal swab samples, researchers can identify tissue-specific expression patterns. This comparison provides a more nuanced understanding of the molecular differences between tissues and may reveal tissue-specific biomarkers for ASD.

eQTL (Expression Quantitative Trait Loci) Analysis

In addition to m-QTL analysis, integrating eQTL (expression quantitative trait loci) analysis will allow the project to identify genetic variants that affect gene expression levels. eQTLs are loci where genetic variations are correlated with changes in gene expression. By analyzing eQTLs, the study can investigate how specific genetic variants influence the transcription of genes related to ASD. This approach helps uncover regulatory pathways and gene networks that contribute to the variability in ASD symptoms. The integration of eQTL analysis with transcriptomic data (such as RNA-Seq) provides a nuanced understanding of how genetic risk factors alter gene expression, ultimately impacting the phenotypic manifestation of ASD.

Epitranscriptomic Analysis

Beyond the study of DNA and RNA through genomics and transcriptomics, epitranscriptomics explores post-transcriptional modifications of RNA, such as N6-methyladenosine (m6A). These RNA modifications can impact mRNA stability, splicing, transport, and translation, thus influencing protein production and cell function. Including epitranscriptomic analysis as part of the RNA-Seq workflow will offer insights into how RNA modifications differ in ASD patients, providing an additional layer of gene regulation that contributes to the complexity of ASD. This investigation could uncover novel epitranscriptomic biomarkers for ASD, adding depth to the study's exploration of gene regulation at the RNA level.

Data Integration and Bioinformatics The integration of the genomic, epigenomic, and transcriptomic data is a key component of the project. The bioinformatics and data analysis teams are responsible for processing and analyzing the vast amounts of data generated by the omics divisions. This involves the use of advanced bioinformatics tools and statistical models to integrate the data and uncover meaningful patterns.

The integrated dataset is subjected to multivariate regression models, which examine the interactions between genetic variants, epigenetic modifications, and gene expression levels. These models are used to identify how these factors jointly contribute to ASD risk and symptom severity. By incorporating both genetic and environmental data, the models can also explore gene-environment interactions that may play a role in the development of ASD.

Network analysis is another key tool used by the bioinformatics team. This technique visualizes the interactions between genes, proteins, and regulatory elements, allowing researchers to identify key genes and pathways that may be involved in ASD. Network analysis also helps to uncover gene regulatory networks that may be disrupted in individuals with ASD, providing insights into the molecular mechanisms that drive the disorder.

The project also leverages machine learning (ML) and artificial intelligence (AI) algorithms to analyze the data. These predictive models are designed to assist clinicians in making personalized treatment decisions based on the molecular profile of each patient. For example, AI models may be used to predict the severity of ASD symptoms based on genetic, epigenetic, and clinical data, allowing for more targeted interventions.

Hi-C and In-Silico Analysis:

While traditional Hi-C analysis often uses crosslinkers to capture long-range chromatin interactions, this project will take a distinct approach by forgoing the use of crosslinkers to link specific DNA fragments. Instead, the chromatin interaction data will be derived and revisited in-silico post-data integration. By analyzing the 3D chromatin architecture computationally, the project will aim to identify spatial chromatin interactions that contribute to the regulation of ASD-associated genes.

This post-integration approach allows for the identification of regulatory elements, such as enhancers and promoters, that interact with distant genomic regions in the context of ASD. The data generated from the genomic, epigenomic, and transcriptomic analyses will be integrated to reveal chromatin interaction patterns that influence gene expression, particularly those associated with ASD pathology. This strategy will allow for a more flexible and refined understanding of 3D genome organization without the limitations imposed by crosslinker-based methods.

ChIP-Seq and In-Silico Epigenetic Pathogenesis Analysis:

In addition to chromatin interaction mapping, ChIP-Seq data will be utilized for epigenetic pathogenesis analysis. By performing in-silico analysis of ChIP-Seq results, the project will identify histone modifications and transcription factor binding sites that are involved in the regulation of gene expression in ASD. This technique will help elucidate the roles of specific epigenetic marks, such as histone acetylation and methylation, in the dysregulation of ASD-associated genes.

The integration of ChIP-Seq data with other omics data, including DNA methylation (WGBS) and RNA-Seq expression profiles, will provide a comprehensive view of the regulatory networks driving ASD. This will allow researchers to pinpoint specific regulatory mechanisms, such as altered transcription factor activity or changes in chromatin accessibility, that may contribute to the onset or severity of ASD symptoms. In-silico analysis of the ChIP-Seq results will thus serve as a powerful tool for understanding the epigenetic landscape associated with ASD pathogenesis.

The project can further enhance its analysis by calculating polygenic risk scores (PRS), which quantify the cumulative effect of numerous small-effect genetic variants on the risk of developing ASD. By aggregating data from thousands of genetic variants, PRS can predict an individual's overall genetic predisposition to ASD. These scores can then be correlated with clinical and phenotypic data to better understand how genetic risk translates into observable symptoms. PRS can also be integrated with environmental and epigenetic data to explore gene-environment interactions, offering a comprehensive model of ASD susceptibility.

Quality Control and Compliance Maintaining the integrity of the project is paramount, and this is achieved through rigorous quality control measures and a comprehensive compliance framework. The project includes several departments dedicated to ensuring that all research activities comply with ethical guidelines and regulatory standards.

The risk management department plays a crucial role in identifying and mitigating potential risks that could compromise the integrity of the study. This department works closely with the internal audit and ethics compliance teams to ensure that all research activities adhere to ethical standards, such as the Helsinki Declaration and national regulations for the protection of personal data.

The quality control teams are responsible for monitoring the quality of the biological samples and ensuring that all data is accurate and reliable. These teams perform regular audits and implement corrective and preventive actions (CAPA) when necessary to address any issues that arise during the course of the study.

The documentation and archiving department is responsible for managing all project records, including audit reports, data transfer logs, and compliance records. This department ensures that all project-related documentation is securely stored and readily accessible for review, facilitating transparency and accountability.

The project also includes a procurement and supply chain management team, which is responsible for ensuring that all necessary materials, equipment, and reagents are procured in a timely manner. This team manages the logistics of material transfers and ensures that all supplies meet the required quality standards.

Ethical Considerations and Participant Safety The safety and privacy of participants are paramount in the conduct of the study. All participant data is anonymized and stored securely to protect their confidentiality. The project adheres to both national and international regulations regarding the protection of personal data, ensuring that participants' rights are respected at all times.

Informed consent is obtained from all participants before they are enrolled in the study. Participants are provided with detailed information about the study's objectives, procedures, and potential risks. They are also informed of their right to withdraw from the study at any time without penalty.

The study has received ethical approval from the relevant national ethics committees, ensuring that all research activities comply with established ethical guidelines. Regular audits are conducted to ensure that all procedures are followed correctly and that any ethical concerns are addressed promptly.

Data Integration and Visualization Upon completion of the study, all data from the genomic, epigenomic, and transcriptomic analyses will be integrated and visualized using state-of-the-art bioinformatics tools. The integrated dataset will provide a comprehensive view of the molecular mechanisms underlying ASD, allowing researchers to identify key biomarkers and potential therapeutic targets.

The integrated data will be presented through various visualization techniques, such as heatmaps, network maps, and pathway diagrams. These visualizations will help researchers interpret the data and draw meaningful conclusions about the biological processes involved in ASD.

Conclusion This project is a landmark study in the field of ASD research, utilizing a multi-omics approach to uncover the genetic, epigenetic, and environmental factors contributing to the disorder. The project's multi-disciplinary structure, with dedicated teams for clinical operations, data analysis, quality control, and compliance, ensures that the research is conducted with the highest level of scientific rigor.

By integrating genomic, epigenomic, and transcriptomic data, the project aims to provide new insights into the molecular mechanisms underlying ASD and to identify potential biomarkers for diagnosis and treatment. The findings from this study could pave the way for personalized medicine approaches to ASD, improving the quality of life for individuals affected by the disorder.

ELIGIBILITY:
- Inclusion Criteria: Autism Spectrum Disorder (ASD) or Autism-like Traits: Individuals diagnosed with ASD based on DSM-5 diagnostic criteria, or those displaying significant autism traits without a formal diagnosis.

Healthy Control Group: Age-, gender-, and socio-demographically matched individuals without any psychiatric or neurological disorder.

ASD Individuals of Varying Functional Levels: Participants with ASD from a broad range of functional abilities, from high-functioning to low-functioning autism.

Comorbid Conditions: Inclusion of volunteers with developmental profiles and comorbid conditions such as ADHD and learning disabilities.

Informed Consent: Written informed consent from participants over 18 years of age. For participants under 18, consent from parents or legal guardians.

- Exclusion Criteria: Severe Psychotic Disorders: Individuals diagnosed with conditions like schizophrenia or schizoaffective disorder.

Known Genetic Syndromes or Chromosomal Anomalies: Individuals with genetic conditions such as Down syndrome or Fragile X syndrome.

History of Genetic or Experimental Therapies: Participants with previous gene or cell therapy, frequent blood transfusions, or bone marrow transplants.

Severe Communication or Cognitive Impairments: Participants with communication or cognitive disorders that would hinder their ability to participate in data collection, or those with aggressive behavioral disorders.

Non-compliance or Medical Restrictions: Individuals unable to comply with study procedures or with medical conditions that prevent biological sample collection.

- Control Group: Healthy Individuals: Participants without ASD or any psychiatric or neurological disorders.

Age and Gender Matching: Matched with the ASD group in terms of age, gender, and socio-demographic status.

No History of Genetic or Neurodevelopmental Disorders: Individuals with no genetic syndromes, chromosomal anomalies, or neurodevelopmental disorders.

No Chronic Disease History: Participants with no history of chronic diseases such as cancer, autoimmune diseases, or metabolic conditions.

Informed Consent: Written informed consent from individuals over 18 years old or from parents/legal guardians for participants under 18.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of individuals diagnosed with Autism Spectrum Disorder (ASD) or exhibiting autism-like traits, selected from clinical centers specializing in neurodevelopmental disorders. The population will also include a healthy control group, matched by age, gender, and socio-demographic variables, recruited from the general community. The ASD cohort will include participants across a range of functional levels, from high-functioning to low-functioning autism, as well as those with developmental profiles and comorbid conditions. Controls will be free of psychiatric or neurological diagnoses and chronic conditions.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2025-12-27 (Estimated); Primary Completion 2027-12-27 (Estimated); Study Completion 2028-05-27 (Estimated)

PRIMARY OUTCOMES:
Finalization of Clinical Data Recruitment | Expected to complete within 24 months of study initiation.
  The primary outcome will be the recruitment of individuals diagnosed with Autism Spectrum Disorder (ASD) and unaffected controls. Comprehensive clinical, sociodemographic, and phenotypic data will be collected, including diagnostic assessments using standardized tools (e.g., ADOS, SCQ).

SECONDARY OUTCOMES:
Collection and Completion of Genetic Raw Data (WGS and WGBS) | Expected to complete within 30 months of study initiation
  he secondary outcome focuses on the acquisition of raw genetic data from whole genome sequencing (WGS) and whole genome bisulfite sequencing (WGBS) from blood and nasal swab samples. The sequencing data will be used for subsequent genetic and epigenetic analyses to identify variants, methylation changes, and their associations with ASD.
Integration of Genetic Data | Expected to complete within 60 months of study initiation.
  This outcome measures the integration of whole genome sequencing (WGS), whole genome bisulfite sequencing (WGBS), and RNA-seq data into a combined dataset for comprehensive multi-omics analysis. The aim is to uncover genetic and epigenetic interactions related to ASD.

OTHER OUTCOMES:
Complete (Final) Outcome Measure : Association Between Clinical and Genetic Data | Expected within 66 months, after all data collection and analysis stages have been completed.
  The final outcome will assess the correlation between genetic, epigenetic, and transcriptomic data with clinical phenotypes. This outcome aims to identify significant associations that may explain the genetic underpinnings of Autism Spectrum Disorder, contributing to potential biomarkers or therapeutic targets.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Torabi, MD.,Ph.D., Study Chair — Selçuk Üniversitesi Tıp Fakültesi Tıbbi Genetik Anabilim Dalı; Ali Kandeğer, MD., Study Director — RUH SAĞLIĞI VE HASTALIKLARI Uzmanı / Konya Selçuk Üniversitesi Tıp Fakültesi- Ruh Sağlığı ve Hastalıkları Anabilim Dalı Anabilim Dalı; Ömer Faruk Akça, MD., Study Director — Çocuk Ve Ergen Ruh Sağlığı Ve Hastalıkları Uzmanı /Konya Necmettin Erbakan Üniversitesi Tıp Fakültesi- Çocuk ve Ergen Ruh Sağlığı ve Hastalıkları Anabilim Dalı; Nadir Koçak, MD, Study Director — Tıbbi Genetik Uzmanı / Konya Selçuk Üniversitesi Tıp Fakültesi- Tıbbi Genetik Anabilim Dalı ve Genetik Hastaliklar Araştırma ve Tedavi Derneği(RTSGD) Yönetim kurulu üyesi; Ebru Marzioğlu Özdemir, MD, Study Director — Tıbbi Genetik Uzmanı / Konya Selçuk Üniversitesi Tıp Fakültesi- Tıbbi Genetik Anabilim Dalı ve Genetik Hastaliklar Araştırma ve Tedavi Derneği(RTSGD) Yönetim kurulu üyesi; Özkan Bağcı, Ph.D., Study Director — Tıbbi Genetik Uzmanı / Konya Selçuk Üniversitesi Tıp Fakültesi- Tıbbi Genetik Anabilim Dalı ve Genetik Hastaliklar Araştırma ve Tedavi Derneği(RTSGD) Yönetim kurulu üyesi
Locations (20):
- Turkey (Türkiye) (20):
  - Konya Selcuk University Faculty of Medicine, Department of Child and Adolescent Psychiatry, Konya, Selçuklu
  - Konya Selcuk University Faculty of Medicine, Department of Psychiatry, Konya, Selçuklu
  - Afyonkarahisar University of Health Sciences, Faculty of Medicine, Department of Child and Adolescent Psychiatry, Afyonkarahisar
  - Ankara Başkent University, Department of Psychiatry, Ankara
  - Ankara Gazi Faculty of Medicine, Department of Child and Adolescent Psychiatry, Ankara
  - Ankara SBÜ Gülhane Faculty of Medicine, Department of Child and Adolescent Psychiatry, Ankara
  - Bursa Uludağ University, Department of Child and Adolescent Psychiatry, Bursa
  - Denizli Pamukkale University Faculty of Medicine, Department of Child and Adolescent Psychiatry, Denizli
  - Erzurum Atatürk University Faculty of Medicine, Department of Child and Adolescent Psychiatry, Erzurum
  - Gaziantep University, Department of Child and Adolescent Psychiatry, Gaziantep
  - Giresun University, Department of Child and Adolescent Psychiatry, Giresun
  - Istanbul Cerrahpasa Faculty of Medicine, Department of Child and Adolescent Psychiatry, Istanbul
  - Istanbul Medeniyet University Faculty of Medicine, Department of Child and Adolescent Psychiatry, Istanbul
  - Istanbul Medeniyet University, Department of Psychiatry, Istanbul
  - Istanbul Çam and Sakura City Hospital, Department of Child and Adolescent Psychiatry, Istanbul
  - Izmir Katip Çelebi Faculty of Medicine, Department of Child and Adolescent Psychiatry, Izmir
  - Konya Necmettin Erbakan University Faculty of Medicine, Department of Child and Adolescent Psychiatry, Konya
  - Konya Selcuk University Faculty of Medicine, Department of Medical Genetics, Konya
  - Şanlıurfa Harran University Faculty of Medicine, Department of Child and Adolescent Psychiatry, Sanliurfa
  - Trabzon Karadeniz Technical University Faculty of Medicine, Department of Child and Adolescent Psychiatry, Trabzon

IPD SHARING:
Plan to Share IPD: Undecided
At this time, the decision to share individual participant data (IPD) has not been finalized. Upon completion of the study, the decision will be reviewed and finalized in accordance with the applicable regulatory and ethical guidelines. The final decision will be subject to obtaining permission from the Turkish Medicines and Medical Devices Agency (TİTCK), the Ethics Committee, and the Turkish Health Ministry. The sharing plan will ensure that all data protection and privacy regulations are strictly followed, and appropriate steps will be taken to safeguard participant confidentiality.

REFERENCES:
- [Background] Trost B, Thiruvahindrapuram B, Chan AJS, Engchuan W, Higginbotham EJ, Howe JL, Loureiro LO, Reuter MS, Roshandel D, Whitney J, Zarrei M, Bookman M, Somerville C, Shaath R, Abdi M, Aliyev E, Patel RV, Nalpathamkalam T, Pellecchia G, Hamdan O, Kaur G, Wang Z, MacDonald JR, Wei J, Sung WWL, Lamoureux S, Hoang N, Selvanayagam T, Deflaux N, Geng M, Ghaffari S, Bates J, Young EJ, Ding Q, Shum C, D'Abate L, Bradley CA, Rutherford A, Aguda V, Apresto B, Chen N, Desai S, Du X, Fong MLY, Pullenayegum S, Samler K, Wang T, Ho K, Paton T, Pereira SL, Herbrick JA, Wintle RF, Fuerth J, Noppornpitak J, Ward H, Magee P, Al Baz A, Kajendirarajah U, Kapadia S, Vlasblom J, Valluri M, Green J, Seifer V, Quirbach M, Rennie O, Kelley E, Masjedi N, Lord C, Szego MJ, Zawati MH, Lang M, Strug LJ, Marshall CR, Costain G, Calli K, Iaboni A, Yusuf A, Ambrozewicz P, Gallagher L, Amaral DG, Brian J, Elsabbagh M, Georgiades S, Messinger DS, Ozonoff S, Sebat J, Sjaarda C, Smith IM, Szatmari P, Zwaigenbaum L, Kushki A, Frazier TW, Vorstman JAS, Fakhro KA, Fernandez BA, Lewis MES, Weksberg R, Fiume M, Yuen RKC, Anagnostou E, Sondheimer N, Glazer D, Hartley DM, Scherer SW. Genomic architecture of autism from comprehensive whole-genome sequence annotation. Cell. 2022 Nov 10;185(23):4409-4427.e18. doi: 10.1016/j.cell.2022.10.009. PMID 36368308
- [Background] Yang C, Sun N, Qin X, Liu Y, Sui M, Zhang Y, Hu Y, Mao Z, Chen X, Mao Y, Shen X. Multi-omics analysis reveals the biosynthesis of flavonoids during the browning process of Malus sieversii explants. Physiol Plant. 2024 Mar-Apr;176(2):e14238. doi: 10.1111/ppl.14238. PMID 38488414
- [Background] Almandil NB, AlSulaiman A, Aldakeel SA, Alkuroud DN, Aljofi HE, Alzahrani S, Al-Mana A, Alfuraih AA, Alabdali M, Alkhamis FA, AbdulAzeez S, Borgio JF. Integration of Transcriptome and Exome Genotyping Identifies Significant Variants with Autism Spectrum Disorder. Pharmaceuticals (Basel). 2022 Jan 27;15(2):158. doi: 10.3390/ph15020158. PMID 35215271
- [Background] Zhou L, Ng HK, Drautz-Moses DI, Schuster SC, Beck S, Kim C, Chambers JC, Loh M. Systematic evaluation of library preparation methods and sequencing platforms for high-throughput whole genome bisulfite sequencing. Sci Rep. 2019 Jul 17;9(1):10383. doi: 10.1038/s41598-019-46875-5. PMID 31316107
- [Background] Bengesser SA, Morkl S, Painold A, Dalkner N, Birner A, Fellendorf FT, Platzer M, Queissner R, Hamm C, Maget A, Pilz R, Rieger A, Wagner-Skacel J, Reininghaus B, Kapfhammer HP, Petek E, Kashofer K, Halwachs B, Holzer P, Waha A, Reininghaus EZ. Epigenetics of the molecular clock and bacterial diversity in bipolar disorder. Psychoneuroendocrinology. 2019 Mar;101:160-166. doi: 10.1016/j.psyneuen.2018.11.009. Epub 2018 Nov 10. PMID 30465968
- [Background] Leontiou CA, Hadjidaniel MD, Mina P, Antoniou P, Ioannides M, Patsalis PC. Bisulfite Conversion of DNA: Performance Comparison of Different Kits and Methylation Quantitation of Epigenetic Biomarkers that Have the Potential to Be Used in Non-Invasive Prenatal Testing. PLoS One. 2015 Aug 6;10(8):e0135058. doi: 10.1371/journal.pone.0135058. eCollection 2015. PMID 26247357
- [Background] Holmes EE, Jung M, Meller S, Leisse A, Sailer V, Zech J, Mengdehl M, Garbe LA, Uhl B, Kristiansen G, Dietrich D. Performance evaluation of kits for bisulfite-conversion of DNA from tissues, cell lines, FFPE tissues, aspirates, lavages, effusions, plasma, serum, and urine. PLoS One. 2014 Apr 3;9(4):e93933. doi: 10.1371/journal.pone.0093933. eCollection 2014. PMID 24699908
- [Background] Xu H, Zhao Y, Liu Z, Zhu W, Zhou Y, Zhao Z. Bisulfite genomic sequencing of DNA from dried blood spot microvolume samples. Forensic Sci Int Genet. 2012 May;6(3):306-9. doi: 10.1016/j.fsigen.2011.06.007. Epub 2011 Jul 6. PMID 21737370
- [Background] Werner B, Yuwono NL, Henry C, Gunther K, Rapkins RW, Ford CE, Warton K. Circulating cell-free DNA from plasma undergoes less fragmentation during bisulfite treatment than genomic DNA due to low molecular weight. PLoS One. 2019 Oct 25;14(10):e0224338. doi: 10.1371/journal.pone.0224338. eCollection 2019. PMID 31652288
- [Background] Hong SR, Shin KJ. Bisulfite-Converted DNA Quantity Evaluation: A Multiplex Quantitative Real-Time PCR System for Evaluation of Bisulfite Conversion. Front Genet. 2021 Feb 25;12:618955. doi: 10.3389/fgene.2021.618955. eCollection 2021. PMID 33719336
- [Background] Chahrour M, O'Roak BJ, Santini E, Samaco RC, Kleiman RJ, Manzini MC. Current Perspectives in Autism Spectrum Disorder: From Genes to Therapy. J Neurosci. 2016 Nov 9;36(45):11402-11410. doi: 10.1523/JNEUROSCI.2335-16.2016. PMID 27911742
- [Background] C Yuen RK, Merico D, Bookman M, L Howe J, Thiruvahindrapuram B, Patel RV, Whitney J, Deflaux N, Bingham J, Wang Z, Pellecchia G, Buchanan JA, Walker S, Marshall CR, Uddin M, Zarrei M, Deneault E, D'Abate L, Chan AJ, Koyanagi S, Paton T, Pereira SL, Hoang N, Engchuan W, Higginbotham EJ, Ho K, Lamoureux S, Li W, MacDonald JR, Nalpathamkalam T, Sung WW, Tsoi FJ, Wei J, Xu L, Tasse AM, Kirby E, Van Etten W, Twigger S, Roberts W, Drmic I, Jilderda S, Modi BM, Kellam B, Szego M, Cytrynbaum C, Weksberg R, Zwaigenbaum L, Woodbury-Smith M, Brian J, Senman L, Iaboni A, Doyle-Thomas K, Thompson A, Chrysler C, Leef J, Savion-Lemieux T, Smith IM, Liu X, Nicolson R, Seifer V, Fedele A, Cook EH, Dager S, Estes A, Gallagher L, Malow BA, Parr JR, Spence SJ, Vorstman J, Frey BJ, Robinson JT, Strug LJ, Fernandez BA, Elsabbagh M, Carter MT, Hallmayer J, Knoppers BM, Anagnostou E, Szatmari P, Ring RH, Glazer D, Pletcher MT, Scherer SW. Whole genome sequencing resource identifies 18 new candidate genes for autism spectrum disorder. Nat Neurosci. 2017 Apr;20(4):602-611. doi: 10.1038/nn.4524. Epub 2017 Mar 6. PMID 28263302
- [Background] Siu MT, Weksberg R. Epigenetics of Autism Spectrum Disorder. Adv Exp Med Biol. 2017;978:63-90. doi: 10.1007/978-3-319-53889-1_4. PMID 28523541
- [Background] Krishnan A, Zhang R, Yao V, Theesfeld CL, Wong AK, Tadych A, Volfovsky N, Packer A, Lash A, Troyanskaya OG. Genome-wide prediction and functional characterization of the genetic basis of autism spectrum disorder. Nat Neurosci. 2016 Nov;19(11):1454-1462. doi: 10.1038/nn.4353. Epub 2016 Aug 1. PMID 27479844
- [Background] Ramaswami G, Won H, Gandal MJ, Haney J, Wang JC, Wong CCY, Sun W, Prabhakar S, Mill J, Geschwind DH. Integrative genomics identifies a convergent molecular subtype that links epigenomic with transcriptomic differences in autism. Nat Commun. 2020 Sep 25;11(1):4873. doi: 10.1038/s41467-020-18526-1. PMID 32978376
- [Background] Gaugler T, Klei L, Sanders SJ, Bodea CA, Goldberg AP, Lee AB, Mahajan M, Manaa D, Pawitan Y, Reichert J, Ripke S, Sandin S, Sklar P, Svantesson O, Reichenberg A, Hultman CM, Devlin B, Roeder K, Buxbaum JD. Most genetic risk for autism resides with common variation. Nat Genet. 2014 Aug;46(8):881-5. doi: 10.1038/ng.3039. Epub 2014 Jul 20. PMID 25038753
- [Background] Geschwind DH, State MW. Gene hunting in autism spectrum disorder: on the path to precision medicine. Lancet Neurol. 2015 Nov;14(11):1109-20. doi: 10.1016/S1474-4422(15)00044-7. Epub 2015 Apr 16. PMID 25891009
- [Background] Sandin S, Lichtenstein P, Kuja-Halkola R, Larsson H, Hultman CM, Reichenberg A. The familial risk of autism. JAMA. 2014 May 7;311(17):1770-7. doi: 10.1001/jama.2014.4144. PMID 24794370
- [Background] Baio J, Wiggins L, Christensen DL, Maenner MJ, Daniels J, Warren Z, Kurzius-Spencer M, Zahorodny W, Robinson Rosenberg C, White T, Durkin MS, Imm P, Nikolaou L, Yeargin-Allsopp M, Lee LC, Harrington R, Lopez M, Fitzgerald RT, Hewitt A, Pettygrove S, Constantino JN, Vehorn A, Shenouda J, Hall-Lande J, Van Naarden Braun K, Dowling NF. Prevalence of Autism Spectrum Disorder Among Children Aged 8 Years - Autism and Developmental Disabilities Monitoring Network, 11 Sites, United States, 2014. MMWR Surveill Summ. 2018 Apr 27;67(6):1-23. doi: 10.15585/mmwr.ss6706a1. PMID 29701730
- [Background] Lord C, Elsabbagh M, Baird G, Veenstra-Vanderweele J. Autism spectrum disorder. Lancet. 2018 Aug 11;392(10146):508-520. doi: 10.1016/S0140-6736(18)31129-2. Epub 2018 Aug 2. PMID 30078460